CLINICAL TRIAL: NCT00770094
Title: A Prospective, Randomized, Multi Center Clinical Comparison Of Fellow Eyes Undergoing Lasik Using The Amo/Visx Customvue™ , The Bausch And Lomb Zyoptix And Planoscan And The Wavelight Allegretto Wave™ Wavefront Guided And Wavefront Optimized Excimer Laser Systems
Brief Title: Multi Laser Platform Comparison Study for LASIK
Acronym: VBLWL-001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Durrie Vision (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Daniel S. Durrie, MD, Durrie Vision
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VBLWL-001
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Myopia; Astigmatism
Keywords: LASIK; Laser Vision correction; Myopia; Myopia with astigmatism; Nearsighted
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Lasers, Excimer; Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment in one eye of the subject and the AMO/VISX CustomVue™ wavefront guided Excimer Laser System performed on the contralateral eye
  Interventions: Device: Excimer Lasers
- Group 2 (Active Comparator): WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment in one eye of the subject and the Bausch and Lomb Zyoptix™ wavefront guided Excimer Laser System performed on the contralateral eye
  Interventions: Device: Excimer Laser for the LASIK procedure
- Group 3 (Active Comparator): WaveLight ALLEGRETTO WAVE™ wavefront optimized excimer laser treatment in one eye of the subject and the Bausch and Lomb Planoscan™ Excimer Laser System performed on the contralateral eye
  Interventions: Device: Excimer Laser for LASIK

INTERVENTIONS:
Device: Excimer Lasers — WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment AMO/VISX CustomVue™ wavefront guided Excimer Laser System
  Arms: Group 1
Device: Excimer Laser for the LASIK procedure — WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment Bausch and Lomb Zyoptix™ wavefront guided Excimer Laser System
  Other Names: LASIK
  Arms: Group 2
Device: Excimer Laser for LASIK — WaveLight ALLEGRETTO WAVE™ wavefront optimized excimer laser treatment Bausch and Lomb Planoscan™ Excimer Laser System
  Other Names: LASIK
  Arms: Group 3

SUMMARY:
Comparison of LASIK outcomes using 3 different lasers and a total of 5 different treatment platforms.

DETAILED DESCRIPTION:
This will be a prospective, randomized, multicenter clinical trial in which up to 180 consecutive eyes scheduled to undergo excimer laser in situ keratomileusis (LASIK) for the correction of myopia with or without astigmatism will be enrolled. Enrolled subjects will have a different Excimer laser system performed in each eye. There will be 30 subjects (60 eyes) in each group.

Group 1: WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment in one eye of the subject and the AMO/VISX CustomVue™ wavefront guided Excimer Laser System performed on the contralateral eye Group 2: WaveLight ALLEGRETTO WAVE™ wavefront guided excimer laser treatment in one eye of the subject and the Bausch and Lomb Zyoptix™ wavefront guided Excimer Laser System performed on the contralateral eye Group 3: WaveLight ALLEGRETTO WAVE™ wavefront optimized excimer laser treatment in one eye of the subject and the Bausch and Lomb Planoscan™ Excimer Laser System performed on the contralateral eye The choice of treatment will first be randomized into one of the three groups and then will also be randomized to the dominant eye prior to LASIK procedure according to the randomization schedule

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have up to -7.00D of spherical equivalent myopia or myopia with astigmatism, with up to -7.00D of spherical component and up to 3.00 D of astigmatic component at the spectacle plane in both eyes.
* Subjects must have a stable refraction as documented by previous clinical records or clinical history. Spherical equivalent has not progressed at a rate of more than 0.50D per year prior to the baseline examination in both eyes or as documented by clinical judgment by the investigator.
* Subjects who wear contact lenses must discontinue wear at least 3 days for soft and at least 3 weeks for RGP prior to the preoperative evaluation or surgery, in either eye.
* Subjects must have visual acuity correctable to at least 20/20 in both eyes.
* Subjects must be at least 18 years of age.
* Subjects must be willing and able to return for scheduled follow up examinations for three months after LASIK surgery.
* Subjects must sign and be given a copy of the written Informed Consent form.

Exclusion Criteria:

* Subjects for whom both eyes do not meet all inclusion criteria and either eye meets any exclusion criteria.
* Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively in either eye.
* Eyes for which the baseline standard manifest refraction exhibits greater than 1.00D more minus in sphere power, or a difference of greater than 0.75 D in cylinder power between eyes.
* Subjects desiring spherical under correction in one eye (i.e. no monovision correction is permitted).
* Subjects for whom the preoperative assessment of the ocular topography and /or aberrations indicates that either eye is not a suitable candidate for LASIK vision correction procedure. Examples include frank or forme frust keratoconus, corneal warpage, and pellucid marginal degeneration, etc.
* Subjects with clinically significant dry eye syndrome or clinically significant blepharitis in either eye.
* Subjects with anterior segment pathology, including clinically significant cataracts or corneal scarring or neovascularization in either eye.
* Subjects with residual, recurrent, active ocular or eyelid disease, including any corneal abnormality (specifically, recurrent corneal erosion, severe basement membrane disease) in either eye.
* Subjects with ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect) in either eye.
* Subjects with unstable (distorted/not clear) corneal mires on central keratometry in either eye.
* Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of surgery for either refractive or therapeutic purposes in either eye.
* Subjects who have a history of Herpes zoster or Herpes simplex keratitis.
* Subjects on chronic systemic corticosteroid or other immunosuppressive therapy that may affect wound healing, any immunocompromised subjects, and subjects with clinically significant atopic disease, connective tissue disease, or diabetes.
* Subjects with a history of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP>23 mm Hg in either eye.
* Subjects with macular pathology in either eye.
* Subjects who are pregnant, lactating, or planning to be pregnant during the course of the study.
* Subjects with known sensitivity to planned study concomitant medications.
* Subjects participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Uncorrected visual acuity | 1 month post operative

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lasik Plus-Galleria, Atlanta, Georgia
  - Lasik Plus Edina, Edina, Minnesota
  - Lasik Plus-Tyson's Corner, McLean, Virginia